CLINICAL TRIAL: NCT07117292
Title: Assessing the Validity and Reliability of Two IMU Sensor Systems and a Goniometer in Multi-Planar Cervical Motion
Brief Title: Assessing the Validity and Reliability of IMU Systems and a Goniometer in Cervical Motion (VIRGO-CM)
Acronym: VIRGO-CM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Collaborators: Brunel University (Other)
Responsible Party: Principal Investigator, George Pamboris, Assistant Professor of Biomechanics and Rehabilitation, European University Cyprus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ΕΕΒΚ ΕΠ 2025.01.231
Record Dates: First submitted 2025-07-22; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cervical Spine Motion Assessment in Healthy Adults
Keywords: Inertial Measurement Units (IMUs); Cervical Spine; Wearable Sensors; Validity; Reliability

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same testing protocol across two sessions. No comparison groups or treatment arms are used. The study involves repeated measures within the same group to assess inter-device validity and intra-device reliability of cervical spine motion measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Sensor-Based Motion Assessment (Experimental): Participants will undergo two testing assessments of cervical spine motion using three devices: Xsens DOT (IMU), Trigno Avanti (IMU), and a universal goniometer. The aim is to assess the validity and reliability of the sensor systems.
  Interventions: Device: Xsens DOT; Device: Trigno Avanti Sensors; Device: Universal Goniometer

INTERVENTIONS:
Device: Xsens DOT — Wearable inertial sensor used to capture cervical range of motion in three planes.
Device: Trigno Avanti Sensors — Wearable inertial sensor used to capture cervical range of motion in three planes.
Device: Universal Goniometer — Standard clinical tool used to measure cervical spine motion angles manually.

SUMMARY:
This study aims to evaluate how accurate and reliable two wearable sensor systems (inertial measurement units or IMUs) and a goniometer are in measuring cervical spine (neck) motion. Healthy adult volunteers will be asked to perform simple head movements in different directions while being assessed using the devices. The goal is to compare how closely these tools agree with each other and how consistently they record motion across repeated tests. This information will help determine whether the sensors are suitable for use in clinical settings to assess neck movement in future patient populations.

DETAILED DESCRIPTION:
This interventional validation study will assess the concurrent validity and test-retest reliability of two inertial measurement unit (IMU) systems (Xsens DOT and Trigno Avanti) and a universal goniometer in measuring multi-planar cervical motion. A within-subject design will be used, with participants performing standardized active cervical range of motion (AROM) tasks in flexion, extension, lateral flexion, and rotation. All measurements will be conducted in a biomechanics lab setting under controlled conditions.

Each participant will undergo three testing sessions:

Familiarization session (optional)

Test session 1

Test session 2

Primary outcomes will include:

Peak angular displacement in each movement plane

Inter-device agreement (validity)

Intra-device test-retest consistency (reliability)

Sensor placement will follow anatomical landmarks based on previous biomechanical research. The IMUs and goniometer will be used simultaneously to compare measurements. Data analysis will involve intraclass correlation coefficients (ICC), standard error of measurement (SEM), and Bland-Altman plots for agreement analysis.

The study will recruit 20-30 healthy adults aged 18-40 with no current or past neck injury. The results will inform future clinical applications of wearable sensors in cervical spine assessment, particularly for populations with neck pain or neuromusculoskeletal disorders.

Ethical approval has been granted by the Cyprus National Bioethics Committee (Approval: ΕΕΒΚ ΕΠ 2025.01.231), and all participants will provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 40 years
* Able to understand and follow instructions
* Provided informed consent

Exclusion Criteria:

* History of cervical spine pathology, trauma, or surgery
* Presence of neck pain, musculoskeletal, neurological, or vestibular disorders
* Use of medications affecting sensorimotor function
* Pregnancy
* Any condition that may interfere with safe participation or data accuracy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Agreement in Cervical Range of Motion between IMUs and Goniometer | Day 1 (single-session assessment)
  Assessment of the validity of two inertial measurement units (Xsens DOT and Trigno Avanti) compared to a universal goniometer in measuring active cervical spine range of motion across flexion/extension, lateral flexion, and axial rotation using Bland-Altman analysis.
Test-Retest Reliability of IMU Systems in Cervical Range of Motion | Day 1 (two repeated assessments within same session)
  Evaluation of intra-session and inter-session test-retest reliability of Xsens DOT and Trigno Avanti inertial sensors in measuring active cervical range of motion (CROM) across three planes (flexion/extension, lateral flexion, rotation). Reliability will be quantified using intraclass correlation coefficients (ICC) and standard error of measurement (SEM).

CONTACTS AND LOCATIONS:
Locations (1):
- European University Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including cervical range of motion measurements and sensor-derived outputs, will be made available upon reasonable request for secondary analysis. Data will be shared via a secure university repository or data-sharing platform following study completion and publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the main findings and will remain accessible for a minimum of 5 years.
Access Criteria: Access to the IPD and supporting materials will be granted to qualified researchers affiliated with academic or research institutions for non-commercial use. Requests should be submitted to the principal investigator and will be evaluated based on the scientific merit of the proposal. Data will be shared via secure transfer through institutional repositories or encrypted platforms.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT07117292/Prot_SAP_000.pdf